CLINICAL TRIAL: NCT03667014
Title: The Impact of Dupilumab on Quality of Life in Moderate to Severe Atopic Dermatitis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dupilimuab Quality of Life
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Atopic Dermatitis; Atopic Dermatitis Eczema
Keywords: atopic dermatitis; eczema; dupilumab
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — dupilumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dupilumab treatment (Experimental): 30 subjects will receive dupilumab for a treatment period of 52 weeks. All patients quality of life measures will be assessed with Psychological General Well-Being scale (PGWB), Work Productivity and Activity Impairment scale (WPAI), and Dermatology Life Quality Index (DLQI). Symptom and satisfaction will be assessed with Treatment Satisfaction Questionnaire for Medication (TSQM), Itch Numerical Rating Scale, Pain Numerical Rating Scale, and Pittsburgh Sleep Quality Assessment (PSQI).
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Dupilumab treatment
  Other Names: Dupixent

SUMMARY:
This is a single-arm, open-label study, which will examine the effect of dupilumab on quality of life in atopic dermatitis patients.

DETAILED DESCRIPTION:
This is a single center, open-label study, which will examine the effect of dupilumab on quality of life in atopic dermatitis (AD). Thirty patients with moderate to severe AD will receive dupilumab for a treatment period of 52 weeks (i.e. last injection on week 48). Improvement in patient quality of life after 52 weeks of treatment with dupilumab will be evaluated using validated dermatologic and non-dermatologic psychometric instruments. The primary endpoint is the improvement in quality of life measured by change in Psychological General Well-Being scale (PGWB) at Week 16 from baseline. Additionally, patients will be given a video recording device to document their experience with the study drug at home. Video footage of patient experiences will be compiled at the end of the study. The compiled video footage will subsequently be watched and analyzed to further understand the experiences of atopic dermatitis patients, and how undergoing dupilumab treatment alters these patients' experiences and attitudes with their skin disease.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with the protocol
* At least 18 years of age
* Diagnosis of atopic dermatitis at least 6 months prior to enrollment, having stable (unchanged) disease for at least 2 months
* Non-immune-compromised status
* Subjects have moderate-to-severe atopic dermatitis, classified as Eczema Area and Severity Index (EASI) score greater than or equal to 6
* Subject is considered a candidate for phototherapy or systemic therapy
* Subjects of child-bearing potential must have a negative urine pregnancy test within 7 days prior to first dose of dupilumab
* Sexually active subjects of childbearing potential must agree to use medically acceptable form of contraception during screening and throughout the study
* Subject meets concomitant medication requirements (see below)

Exclusion Criteria:

* Younger than 18 years of age
* Has mild atopic dermatitis, classified as EASI score less than 6
* History of known or suspected intolerance to any of the ingredients of the investigational study product
* Evidence of skin conditions other than atopic dermatitis that would interfere with study-related evaluations of atopic dermatitis.
* History of immune-compromised status [e.g. human immunodeficiency virus (HIV) positive status or other immune suppressing drug] or a congenital or acquired immunodeficiency or subject testing positive for HIV during screening procedures
* Has a poorly controlled medical condition including, but not limited to, unstable cardiovascular disease, poorly controlled diabetes, recent stroke, history of recurrent infections, or any other condition for which, in the opinion of the investigator, participation in the study would place the subject at risk
* Has a history of or ongoing drug or alcohol abuse
* Is not willing to comply with concomitant medication requirements
* Is known, or suspected of being unable to comply with the study protocol
* Subjects who are well controlled on current treatment for atopic dermatitis and participation in the study may worsen disease control significantly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina Bhutani, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Psoriasis and Skin Treatment Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrouk M, Nakamura M, Zhu TH, Farahnik B, Koo J, Bhutani T. The impact of PASI 75 and PASI 90 on quality of life in moderate to severe psoriasis patients. J Dermatolog Treat. 2017 Sep;28(6):488-491. doi: 10.1080/09546634.2016.1278198. Epub 2017 Jan 18. PMID 28042711
- [Background] Drucker AM, Wang AR, Qureshi AA. Research Gaps in Quality of Life and Economic Burden of Atopic Dermatitis: The National Eczema Association Burden of Disease Audit. JAMA Dermatol. 2016 Aug 1;152(8):873-4. doi: 10.1001/jamadermatol.2016.1978. No abstract available. PMID 27305113
- [Background] Nicholas MN, Gooderham MJ. Atopic Dermatitis, Depression, and Suicidality. J Cutan Med Surg. 2017 May/Jun;21(3):237-242. doi: 10.1177/1203475416685078. Epub 2017 Jan 9. PMID 28300443
- [Background] Sidbury R, Khorsand K. Evolving Concepts in Atopic Dermatitis. Curr Allergy Asthma Rep. 2017 Jul;17(7):42. doi: 10.1007/s11882-017-0710-5. PMID 28555328
- [Background] Simpson EL. Dupilumab Improves General Health-Related Quality-of-Life in Patients with Moderate-to-Severe Atopic Dermatitis: Pooled Results from Two Randomized, Controlled Phase 3 Clinical Trials. Dermatol Ther (Heidelb). 2017 Jun;7(2):243-248. doi: 10.1007/s13555-017-0181-6. Epub 2017 May 13. PMID 28503712

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Additional participants were recruited due to high number of dropouts related to the COVID19 pandemic
Groups:
- Dupilumab Treatment: 34 subjects will receive dupilumab for a treatment period of 52 weeks. All patients quality of life measures will be assessed with Psychological General Well-Being scale (PGWB), Work Productivity and Activity Impairment scale (WPAI), and Dermatology Life Quality Index (DLQI). Symptom and satisfaction will be assessed with Treatment Satisfaction Questionnaire for Medication (TSQM), Itch Numerical Rating Scale, Pain Numerical Rating Scale, and Pittsburgh Sleep Quality Assessment (PSQI).
  Dupilumab: Dupilumab treatment
Period: Overall Study
Arm/Group | Dupilumab Treatment
Started | 34
Completed | 24
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Dupilumab Treatment
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 17
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 12
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Psychological General Well-Being Scale (PGWB)
Description: The primary endpoint is the improvement in quality of life measured by change in Psychological General Well-Being scale (PGWB) at Week 16 from baseline. It is a self-reported, 22 item questionnaire, scored 0-5 and summed. PGWB will be administered at every study visit.
Time Frame: 16 weeks
Population: All patients completing 52 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab Treatment
Number analyzed (Participants) | 24
score on a scale
  Baseline | 68.3 (19.5)
  Week 16 | 73.7 (23.7)

2. Secondary Outcome: Work Productivity and Activity Impairment Scale (WPAI:SHP)
Description: Improvement in work productivity measured by change in Work Productivity and Activity Impairment scale (WPAI) at Week 16 from baseline. It measures the effect of health and symptom severity on work productivity and nonwork activities by assessing absenteeism, presenteeism, and impairment of daily activities. There are 6 questions, each with unique answers. WPAI outcomes are expressed as impairment percentages (0-100), with higher numbers indicating greater impairment and less productivity.
  Scoring equations:
  1. Percent work time missed due to problem: Q2/(Q2+Q4)
  2. Percent impairment while working due to problem: Q5/10
  3. Percent overall work impairment due to problem:
     Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4)))x(Q5/10)]
  4. Percent activity impairment due to problem: Q6/10
Time Frame: 16 weeks
Population: 24 patients who completed 52 weeks of the study
Measure: Mean (Standard Deviation); unit: percentage of overall work impairment
Arm/Group | Dupilumab Treatment
Number analyzed (Participants) | 24
percentage of overall work impairment
  Baseline | 0.45 (0.26)
  Week 16 | 0.24 (0.25)

3. Secondary Outcome: Dermatology Life Quality Index (DLQI)
Description: Improvement in quality of life measured by change in Dermatology Life Quality Index (DLQI) at Week 16 from baseline. It is a 10 item questionnaire with a final score calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Time Frame: 16 weeks
Population: 24 subjects completing 52 weeks of study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab Treatment
Number analyzed (Participants) | 24
score on a scale
  Baseline | 16.4 (7.0)
  Week 16 | 8.0 (6.8)

4. Secondary Outcome: Itch Numerical Rating Scale
Description: Improvement in itch scores using numerical rating scales at Week 16 from baseline. This is a 0-10 scale with 0 equaling No itch, and 10 being Worst imaginable itch. Patients will circle number that describes the itch experienced from atopic dermatitis.
Time Frame: 16 weeks
Population: 24 subjects completing 52 weeks of the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab Treatment
Number analyzed (Participants) | 24
score on a scale
  Baseline | 7.7 (2.0)
  Week 16 | 3.5 (2.6)

5. Secondary Outcome: Pain Numerical Rating Scale
Description: Improvement in pain scores using numerical rating scales at Week 16 from baseline. This is a 0-10 numerical scale with 10 as the worst imaginable itch. Patients circle the number that best describes the pain experienced from atopic dermatitis.
Time Frame: 16 weeks
Population: 24 subjects completing 52 weeks of the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab Treatment
Number analyzed (Participants) | 24
score on a scale
  Baseline | 5.3 (3.2)
  Week 16 | 2.0 (2.3)

6. Secondary Outcome: PSQI
Description: Improvement in sleep quality measured by the Pittsburgh Sleep Quality Assessment (PSQI) at Week 16 from baseline. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Time Frame: 16 weeks
Population: 24 patients who completed 52 weeks of study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab Treatment
Number analyzed (Participants) | 24
score on a scale
  Baseline | 10.05 (4.58)
  Week 16 | 6.59 (4.38)

ADVERSE EVENTS:
Time Frame: 52 Weeks
Arm/Group | Dupilumab Treatment
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 3/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dupilumab Treatment (N=34)
Facial erythema (Skin and subcutaneous tissue disorders) | 1
Eye redness (Skin and subcutaneous tissue disorders) | 1
Eyelid swelling (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT03667014/Prot_SAP_000.pdf